CLINICAL TRIAL: NCT01722838
Title: An Evaluation of a Locally Developed Homegrown HIV Prevention Intervention
Brief Title: Black Men Evolving Behavioral HIV Prevention Intervention for Black MSM
Acronym: B-ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5U01PS001574 (NIH); PS09-007 (Other: CDC/DHAP)
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: HIV CDC Category A1
Keywords: Black MSM; HIV Prevention

STUDY DESIGN:
Intervention Model Description: Assignment to behavioral intervention or comparison group
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B-ME intervention (Experimental): Men will receive behavioral HIV prevention intervention, B-ME.
  Interventions: Behavioral: B-ME Intervention
- Control Arm (No Intervention): Men in this arm will receive monthly text or telephone voice messages relaying general health messages.

INTERVENTIONS:
Behavioral: B-ME Intervention — B-ME is a behavioral intervention of HIV prevention risk reduction administered in a group format during a 2.5 day retreat (19 hours) format.
  Arms: B-ME intervention

SUMMARY:
B-ME is a research intervention study designed to address the needs of African American men who have sex with men (AAMSM) who are at high risk for HIV. The intent of the intervention is to decrease HIV risk behaviors among African American MSM using an intervention developed by and for African American MSM.

The hypothesis guiding this study is: that participants who complete B-ME intervention will report greater reductions in sexual risk behaviors than the standard of care comparison group.

DETAILED DESCRIPTION:
The Specific Aims of this study are 1) to further explicate and develop the intervention, 2) to evaluate its efficacy in reducing HIV risk behaviors and 3) to expand the limited body of research on HIV prevention/risk reduction practices for African American men who have sex with men(AAMSM). The study will use a randomized-controlled trial design to compare receiving B-ME intervention to receiving basic men's health and wellness messaging (standard of care), hypothesizing: hypothesizing: that participants who complete B-ME intervention will report greater reductions in sexual risk behaviors than the standard of care comparison group. The study will utilize a pre-test/post-test design with participants randomized to intervention and comparison groups; have a strategy to retain at least 80% of participants through study completion; collect data at baseline, at 3 months post-intervention, and at 6 months post-intervention; and rigorously measure outcomes that directly impact HIV risk. Data will be collected at each assessment point to assess B-ME's ability to improve behavioral outcomes that directly impact Black MSM HIV risk: (1) number of unprotected anal and vaginal sex events; (2) number of unprotected sex events with persons of unknown HIV status; (3) frequency of HIV testing, and (4) increased communication between partners about sex and strategies for reducing the risk of HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* a) Be 18 to 55 years old b) Self identify as African American (Black national) c) Self identify as a male (because this is a study of an intervention to impact change among Black MSM, only self identified males will be included, therefore no females or transgendered identified persons will be included).

  d) Report being sexually active in the past 30 days (ie., one or more instances of vaginal or anal sex with a male or female) e) Report at least one instance of unprotected anal or oral sex with a male identified partner in the past year f) Have not previously participated in the CTCA intervention. g) Have not received an evidence-based HIV prevention intervention in the past 180 days

Exclusion Criteria:

* Men are ineligible to participate in the trial if they:

  1. Identify as a transgender woman; OR
  2. Plan to move before the end of the study; OR
  3. Have participated in any HIV or substance use prevention studies in the last 180 days.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 438 (Actual)
Dates: Start 2012-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
reductions in sexual risk behaviors | baseline, 3-month, 6-month
  Unprotected anal or vaginal sex and condom use during

CONTACTS AND LOCATIONS:
Overall Officials: Darrell P Wheeler, PHD MPH, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Chicago, Chicago, Illinois, United States